CLINICAL TRIAL: NCT01836094
Title: Beneficial Effects of Methylene Blue on Human Cognitive and fMRI Measures
Brief Title: Effects of USP Methylene Blue on Cognitive and fMRI Brain Activity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: NS 13-208
Record Dates: First submitted 2013-04-12; First posted 2013-04-19 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Brain Activity
Keywords: Methylene Blue; Memory; Mental Fatigue; Brain metabolism; fMRI; psychomotor vigilance task (PVT); delayed match-to-sample memory task; PVT; DMS
MeSH Terms: conditions — Mental Fatigue | interventions — Methylene Blue; Indigo Carmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylene Blue (Experimental): Methylene Blue, 280mg, oral, one time
  Interventions: Drug: Methylene Blue (USP grade, 280mg oral)
- Placebo (Placebo Comparator): FD&C Blue No. 2 (food dye), oral, one time
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylene Blue (USP grade, 280mg oral)
  Other Names: USP Methylene Blue, Phenothiazin-5-ium, 3, 7-bis (dimethylamino)-chloride, trihydrate
  Arms: Methylene Blue
Drug: Placebo — oral, one time
  Other Names: FD&C Blue No. 2 (food dye)
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether low-dose USP methylene blue (MB) will: i) improve short-term memory retention in a delayed match-to-sample task, ii) reduce reaction time in a psychomotor vigilance test, and iii) enhance responses to a visual-motor task as measured by functional magnetic resonance imaging (fMRI).

A single low-dose MB or placebo will be orally administered to self-declared healthy adults using double-blind study design. Non-invasive fMRI data will be acquired before and after MB administration in the same subjects. Each study will take 2-3 hours, inclusive of an hour break in between.

DETAILED DESCRIPTION:
Self-declared healthy adult volunteers will be studied using a double-blind, placebo-controlled design. After informed consent and familiarity with the tasks and the MRI environment, the subject will enter an MRI scanner and perform the following 3 tasks:

Delayed match-to-sample task: The subject views an object for a few seconds. After a few (variable) seconds, the subject is presented with two patterns and the subject needs to press the left or right button based on whether the picture on the left or the right is the same as the previous picture. The correct and incorrect answers are recorded. A few of these trials will be cycled, lasting about 5-10 mins.

Psychomotor vigilance test: The subject will receive a visual cue to press a button as fast as possible. The reaction time is recorded. A false start is when the subject presses before the visual cue and that trial is not counted. The subject is instructed to avoid a false start. A few of these trials will be cycled, lasting about 5-10 mins.

Visual-motor task: The subject is instructed to tap his/her 4 fingers against the thumb every second and cycle through the 4 fingers, in synchrony with an alternating visual checkerboard patterns. A few of these trials will be cycled, lasting about 5-10 mins.

For calibration of the fMRI signal, fMRI data will also be acquired during a brief (3-5 mins) inhalation of 5% CO2 in air.

fMRI measurements will be made before intervention. The subject comes out of the scanner, orally ingests the USP MB or placebo, and waits for an hour (break). The same measurements will then be repeated.

fMRI data acquisition: The MRI pulse sequences include standard and non-invasive anatomical MRI for co-registration, blood flow and blood-oxygen-level dependent (BOLD) fMRI. fMRI will image changes in regional brain activity associated with these tasks.

In addition, one week after the fMRI study, the subject will be emailed a short questionnaire (which takes a few minutes to answer) and the responses can be returned via email.

Data analysis: Standard fMRI analysis will be analyzed using established fMRI software. Statistical parametric analysis will be performed to generate activation maps. Task-evoked changes in brain activities will be analyzed and contrasted between placebo and MB conditions in the same subjects. Paired t-test will be used for group comparison with P < 0.05 (with bonferroni correction) considered statistically significant.

Expected results: The investigators predict that, compared to placebo, MB will: i) improve short-term memory retention in a delayed match-to-sample task by memory performance and enhanced fMRI responses in the prefrontal cortex-hippocampus, ii) reduce reaction time in a psychomotor vigilance test and enhanced fMRI responses within a cortical sustained attention network and the motor systems, and iii) enhance responses in the visual and motor cortices.

Power analysis: Sample sizes were calculated for a power of 80%, alpha = 0.05 to detect statistical difference between MB and placebo. The investigators estimate they will need 40 subjects (complete studies) and thus will recruit 50 subjects to account for potential failed studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years, self declared healthy individuals
* English speaker and be able to give consent

Exclusion Criteria:

* Contraindication for MRI (pacemaker, metal implants, etc.)
* Claustrophobia
* Pregnant (child-bearing age females will be tested to exclude pregnancy onsite)
* Breast-feeding
* A history of hypersensitivity or allergy to methylene blue, glucose-6-phosphate dehydrogenase deficiency (determined via questionnaire)
* Neurological, mental, or cardiovascular disorders
* Liver, kidney disorders, kidney or liver transplant, hypertension, diabetes, etc.
* Known hypersensitivity to thiazide diuretics and phenothiazines
* A history of a psychotic disorder or panic disorder, violent or suicidal behavior, psychiatric institutionalization or imprisonment
* Any other condition, which in the opinion of the investigator, would put the participant at risk and warrant exclusion from the study
* Methemoglobinemia
* On any psychiatric serotonergic antidepressant medication or drugs of abuse currently or within the last 5 weeks
* History of panic attack
* Color Blindness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Improvement in reaction time assessed by fMRI measurements and PVT measurements | 1 hour
  fMRI will be assessed using standard fMRI analysis tools. Psychomotor-Vigilance-Test (PVT) measurements will be made using a computer program written in Psychology Experiment Building Language (PBL).
Improvement in memory assessed by fMRI measurements and DMS measurements | 1 hour
  fMRI will be assessed using standard fMRI analysis tools. Delayed-match-to-sample task (DMS) measurements will be made using a computer program written in Psychology Experiment Building Language (PBL).

SECONDARY OUTCOMES:
Enhanced fMRI responses to visual-motor task | 1-2 hours
  fMRI will be assessed using standard fMRI analysis tools.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Q. Duong, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Research Imaging Institute, The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Background] Riha PD, Bruchey AK, Echevarria DJ, Gonzalez-Lima F. Memory facilitation by methylene blue: dose-dependent effect on behavior and brain oxygen consumption. Eur J Pharmacol. 2005 Mar 28;511(2-3):151-8. doi: 10.1016/j.ejphar.2005.02.001. PMID 15792783
- [Background] Gonzalez-Lima F, Bruchey AK. Extinction memory improvement by the metabolic enhancer methylene blue. Learn Mem. 2004 Sep-Oct;11(5):633-40. doi: 10.1101/lm.82404. PMID 15466319
- [Background] Wrubel KM, Riha PD, Maldonado MA, McCollum D, Gonzalez-Lima F. The brain metabolic enhancer methylene blue improves discrimination learning in rats. Pharmacol Biochem Behav. 2007 Apr;86(4):712-7. doi: 10.1016/j.pbb.2007.02.018. Epub 2007 Mar 6. PMID 17428524
- [Background] Wen Y, Li W, Poteet EC, Xie L, Tan C, Yan LJ, Ju X, Liu R, Qian H, Marvin MA, Goldberg MS, She H, Mao Z, Simpkins JW, Yang SH. Alternative mitochondrial electron transfer as a novel strategy for neuroprotection. J Biol Chem. 2011 May 6;286(18):16504-15. doi: 10.1074/jbc.M110.208447. Epub 2011 Mar 18. PMID 21454572
- [Background] Lim J, Wu WC, Wang J, Detre JA, Dinges DF, Rao H. Imaging brain fatigue from sustained mental workload: an ASL perfusion study of the time-on-task effect. Neuroimage. 2010 Feb 15;49(4):3426-35. doi: 10.1016/j.neuroimage.2009.11.020. Epub 2009 Nov 24. PMID 19925871
- [Background] Bruchey AK, Gonzalez-Lima F. Behavioral, Physiological and Biochemical Hormetic Responses to the Autoxidizable Dye Methylene Blue. Am J Pharmacol Toxicol. 2008 Jan 1;3(1):72-79. doi: 10.3844/ajptsp.2008.72.79. PMID 20463863